# Notification of the second interim analysis of a clinical trial or of a research project BASEC 2019-00646 (24 May 2022)

# 1. General study information

| BASEC or PB_BASEC ID number | 2019-00646; ClinicalTrials.gov NCT0404830 |
|---|---|
| Title of the study | Short postsurgical antibiotic therapy for spinal infections: protocol of prospective, randomized unblinded, noninferiority trials (SASI trials). |
| Lead Ethics Committee (Swiss EC only) | Zurich |
| Sponsor | Prof. Dr. med. Ilker Uçkay |
| Principal Investigator | PD Dr. med. Michael Betz |
| Was the study carried out in other countries than Switzerland? | Yes No X (Swiss study only) |
| International protocol publication | Betz M, Uçkay I, Schüpbach R, Gröber T, Botter SM, Burkhard J, Holy D, Achermann Y, Farshad M. Short postsurgical antibiotic therapy for spinal infections: protocol of prospective, randomized, unblinded, noninferiority trials (SASI trials). Trials. 2020 Feb 6;21(1):144. doi: 10.1186/s13063-020-4047-3. |
| | According to the study protocol, three interim analyses are foreseen: after the inclusion of the first 20, 60, and 120 patients. The results of the first interim analysis after 20 testing episodes have been presented internally. |
| Context of this 2 <sup>nd</sup> interim analysis | Now, with 50 episodes complete and 48 further episodes on way, we anticipate the second interim analysis from the first 60 to the 50 completed cases. Additionally, the writing of this analysis coincidences with the 2 <sup>nd</sup> anniversary of the study start. We write this second interim analysis in the form of a report |
| Date of 2 <sup>nd</sup> interim analysis | 31 July 2021 |

| Approval by the independent study data committee | 24 May 2022 |
|--------------------------------------------------|-------------|

## 2. Early termination

| Has the study been terminated prematurely? | No | X go to section 3. Study duration |
|---|---|---|
|---|---|---|

## 3. Study duration

| Date: Study start in Switzerland Study involving persons: Date first patient/ first visit in Switzerland. Study not involving people: data/sample collection started. | 7 August 2019 |
|---|---|
| <ul> <li>Date: End of study in Switzerland</li> <li>Study involving persons: Date last patient / last visit in Switzerland.</li> <li>Study not involving persons: data/sample collection completed.</li> </ul> | ongoing |
| Study completed? | Yes ☐ No ☒ N/A (Swiss study only) |

## 4. Details on participating center(s)

| Number of participating center(s) in Switzerland | |
|---|---|
| Active open center(s): 2 | Balgrist University Hospital; Zollikerberg Hospital |

## 5. Details on recruitment

| Number of participants in Switzerland | | | |
|---|---|---|---|
| Target number: 236 | Enrolled:<br>100 | Prematurely terminated (drop-outs): | Completed<br>(end-of<br>treatment)<br>50 |

If possible, explain any gap between target number and enrolled number of participants

Study ongoing with the half of the patients not having finished the minimal follow-up period, few dropouts

#### 6. Final study report (clinical trials only)

| | Yes |
|---|---|
| Is a summary of the final report on the clinical trial available and enclosed with this form? | No Signature If No, submit to the (Lead-) Ethics Committee within a year after completion or discontinuation of the clinical trial. |

#### 7. Interim results, absence of major biases and provisory non-inferiority assessments

Briefly, the trials involves two strata of operates spine infections: with and without remaining infected osteosynthesis material. The 1:1 randomisation allocates half of the eligible patients into a short and a long postoperative antibiotic arm; which are 3 vs. 6 weeks in absence of a residual infected implant; or 6 vs. 12 weeks in case of a remaining infected implant. The study target are 236 infection episodes and non-inferiority is set at a margin of 10%. The minimal follow-up for implant-related infections is 1 year.

#### 7.1. No major inclusion bias

Of 170 potentially eligible patients, 96 (56%) have been included in the study. The population of included and excluded patients are similar regarding key elements of spine infections. The sex, the median number of surgical debridement, the presence of an infected implant, as well as the proportion of key pathogen such as *S. aureus* or Gram-negative germs did not differ between the included and the excluded infections. The only important difference is that excluded patients are treated longer with systemic antibiotics, which is the *raison d'être* of this trial. In other words, participation in these SASI trials reduced the overall duration of antibiotic prescription among the spine infection patients.

## 7.2. Clinical failures and microbiologically-identical recurrences

The number of clinical failures after the end of treatment are 4 (4/96; 4%), of which two are true microbiological recurrence due to *S. aureus*; occurring in the same patient, who is a formed IV drug addict patient. The other two failures are a secondary endocarditis during treatment and clinical failure without the proof of recurrent pathogens. The number of failures are small and better than most literature reporting the outcome of spine infections.

| Intention-To-Treat population | Short antibiotic arm | Long antibiotic arm |
|---|---|---|
| Failures implant-related infections | 2/31 | 0/31 |
| Failures non-implant infections | 1/15 | 1/19 |
| - of which microbiological recurrences | 1/15 | 1/19 |

#### 7.3. Adverse events

The number of mild, moderate and severe adverse events were equally distributed between the short and long antibiotic arms. For implant-free spine infections, these proportions were 47% vs. 41%. They



Schweizerische Ethikkommissionen für die Forschung am Menschen Commissions d'éthique suisses relative à la recherche sur l'être humain Commissioni etiche svizzere per la ricerca sull'essere umano Swiss Ethics Committees on research involving humans

were 65% vs. 71% for implant-related infections, when including the mild events. Among all 59 single adverse events, 36 (61%) yielded a link to the antibiotic treatment of various extent. Most adverse events occurred within three weeks of therapy start. The corresponding differences between the short and long antibiotic arms were all insignificant.

| Fatal cases: | Serious Adverse<br>Events (SAEs): | | us Adverse Drug<br>ions SADRs | Suspected Unexpected<br>Serious Adverse Reactions,<br>0 |
|---|---|---|---|---|
| Have all safety cases been reported to the (Lead-) Ethics Committee within the regulatory timelines? | | Yes | $\boxtimes$ | |
| | | No | | |
| | | N/A | | |

### 7.4. Non-inferiority assessments

In the ultimate Per-Protocol population analysis, and solely for implant-related infections, so far only the outcome "microbiologically-confirmed infectious recurrence" fulfils the statistical non-inferiority requirements (5.6% percentage points [90%Cl 9.2% to 9.8%]). Regarding the overall clinical failures or the stratum of implant-free spine infections, the calculations with the available study populations are underpowered. They cannot be definitively assessed by now due to (yet) insufficient follow-up times.

## 8. Signature of the applicant

I hereby confirm that / confirm that (

The above information given on this declaration is correct; and

J. W.S

Date and place: Zurich, 24 May 2022

**Print names:** Prof. Dr. med. Ilker UCKAY; PD Dr. med. Michael Betz

Signatures: